CLINICAL TRIAL: NCT02547298
Title: Correlation Between Urinary Symptoms and Interstitial Cystitis (IC)-Like Findings on Cystoscopy With Hydrodistension
Brief Title: Interstitial Cystitis (IC)-Like Findings With Hydrodistension
Status: Terminated | Type: Observational
Why Stopped: Previous PI left, staffing changes especially in setting of COVID pandemic meant we no longer wanted to proceed with further recruitment. There were no adverse events or concerns leading to the termination of the study. Simply logistical concerns
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Ioana Marcu, MD, MD, St. Louis University
Other Study IDs: 25534
Record Dates: First submitted 2015-08-26; First posted 2015-09-11 (Estimated); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: All participants will be filling out questionnaires and undergoing cystoscopy with hydrodistension for evaluative reasons

SUMMARY:
Patients who are already scheduled to have a gynecologic, urologic or uro-gynecologic procedure involving cystoscopy (a lighted scope is used to look inside the bladder) under anesthesia will be approached to participate in the study. Once prospective study subjects are consented, they will be requested to complete the study questionnaires.

At the time of the procedure, during the cystoscopy, patients will undergo hydrodistension (stretching the bladder with fluid). Photographic images of the bladder will be collected, to be later analyzed by examiners. Patients who have positive findings for interstitial cystitis during cystoscopy with hydrodistension, will be notified of the findings after the procedure.

They will be asked to fill out an additional, previously completed questionnaire at the time of a follow-up visit, during a phone interview or responding to the questionnaire via a secure web site. These patients will be treated for interstitial cystitis by their primary providers as clinically indicated.

DETAILED DESCRIPTION:
Patients who are already scheduled to have a gynecologic, urologic or uro-gynecologic procedure involving cystoscopy will be approached to participate in the study. They will be approached either at the time of an office visit or on the day of the scheduled procedure in the preoperative area.

Study-Related Once consented, they will be requested to fill out the study questionnaires. IC Problem Index/IC symptom Index, Pelvic Pain and Urgency/Frequency Patient Symptom Scale(PUF), IBS (Irritable Bowel Syndrome) questionnaire, Functional Esophageal Disorder Questionnaire, and Painful Bladder questionnaire. Completion of these questionnaires should take approximately 15 minutes.

All patients will undergo cystoscopy with hydrodistension as part of the study protocol. Cystoscopy with hydrodistension is used as a diagnostics/evaluative test.

Cystoscopy-Standard of care The bladder will be be emptied prior to cystoscopy. Cystoscopy will be performed with a 5 mm 30o or 70o cystoscope. The angle of view through the scope (or what the physician sees) is described as 30 degrees or 70 degrees. Sterile saline or water will be infused under direct visualization. Fluid bag will be held at 80 cm above the patient. After 200 cc's of filling the infusion will be stopped. This is the standard procedure for cystoscopy. A resurvey of the bladder will be performed. A minimum of two pictures will be taken - one of the back wall and one of the dome of the bladder. Any abnormal findings will be recorded as well.

Hydrodistension- standard of care or study related. The bladder will be filled by gravity (no pressure) the fluid bag is held 80-100cm above the bed level and the bladder is filled by gravity. Fluid will stop when the bladder reaches capacity or the physician will stop the flow when 700cc is reached. Once the bladder is filled, it is then partially emptied. This procedure should take no more than 60 seconds. The bladder is left partially filled so the physician can take a final look (resurvey) at the bladder before the procedure is completed and the scope withdrawn. This is the standard procedure for hydrodistension. At least five pictures will be taken: trigon, left and right bladder wall, posterior wall of the bladder, and dome of the bladder. A short video clip (approximately 10-15 seconds long) will be taken as well for documentation. Again, any abnormal findings will be documented.

Image review-study related Cystoscopic images will be de-identified and pooled. Batches of 25 sets of images will be evaluated by a panel of urogynecologists. Each reviewer will evaluate each set of images, ranking them as: positive, equivocal or negative for interstitial cystitis findings. A minimum of 10 glomerulations per quadrant in 3 out of 4 quadrants, or any Hunner ulcers will be required for positive diagnosis. Glomerulations will be graded by distribution and number. Additional findings will be recorded: trabeculations, metaplasia, masses, stones, etc. In cases of equivocal findings, the panel can review video clip that may contain additional visual information.

Study related Patients who have positive findings for interstitial cystitis during cystoscopy with hydrodistension, will be notified of the findings after the procedure. At their 4 week and 6 month followup visits these patients will be asked to fill out the IC Problem Index/IC symptom Index questionnaire, this will be compared to the same questionnaire the patient filled out pre op. If the patient is unable to come to the office they may receive a phone call to complete the questionnaire or if they have access to e-mail they may be able to complete the questionnaire on a secure web base site (Red Cap). The follow up questionnaire will not be completed by those who are not diagnosed with interstitial cystitis and their participation in this study will end after the procedure, and they will be referred back to their primary or referring physician for follow up.

Study related The patient's medical record will also be reviewed for history and demographics.

Standard of care Patients with IC will be treated by their primary providers as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Patients must be at least 18 years of age.
3. Patients must have been previously scheduled for a surgical procedure that includes cystoscopy under anesthesia or cystoscopy with hydrodistension under anesthesia.
4. Patients must be able to provide written informed consent.

Exclusion Criteria:

1. pregnancy
2. planned cystotomy
3. incidental cystotomy during surgery - patient not eligible for hydrodistention
4. patient's age > 90
5. history of pelvic radiation 6, Previous or newly diagnosed bladder tumor

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women scheduled to undergo cystoscopy or cystoscopy with hydrodistension in an academic institution, within the benign gynecologic division with eligibility criteria as above.
Sampling Method: Probability Sample
Enrollment: 734 (Actual)
Dates: Start 2015-06; Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Correlation between severity of urinary symptoms and IC-like findings on cystoscopy with hydrodistension. | up to 5 years
  Change From Baseline in Pain on the 11 point Short Pain Scale (SPS-11).

SECONDARY OUTCOMES:
The association of GI symptoms with IC-like findings on cystoscopy with hydrodistension | up to 5 years
  Correlation between questionnaires responses and cystoscopic findings
The correlation between O'Leary-Sant score and cystoscopic findings | up to 5 years
  correlation between O'Leary-Sant score and cystoscopic findings
The correlation between PUF score and cystoscopic findings | up to 5 years
  Correlation between PUF score and cystoscopic findings
The association between cystoscopic and previous urologic or gynecologic surgeries | up to 5 years
  Correlation between cystoscopic and previous urologic or gynecologic surgeries
The number of patients with interstitial cystitis who's symptoms improve after cystoscopy with hydrodistension | up to 5 years
  To evaluate the number of patients with interstitial cystitis who's symptoms improve after cystoscopy with hydrodistension based on questionnaire responses
Cystoscopic findings in this patient population | up to 5 years
  To evaluate other cystoscopic findings in this patient population based on review of reports and photos
The safety and complications after cystoscopy with hydrodistension | up to 5 years
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Ioana Marcu, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No